CLINICAL TRIAL: NCT05177627
Title: Integrating the Fundamentals of Care Framework Into Italian Nursing Education
Acronym: FoC-FORM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Milko Zanini, Assistant Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FoC-FORM 2021
Record Dates: First submitted 2021-10-13; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Nursing Students

STUDY DESIGN:
Intervention Model Description: Students participating in the study will be randomly assigned to two groups:
  1. experimental group with educational interventions of integration of the FoC framework (learning according to the FoC framework with the contents of the current curriculum);
  2. control group without intervention (learning according to the current educational model and the contents of the current curriculum); A researcher not involved in the educational interventions and data collection of the study at the University of Genoa will randomly assign in a 1: 1 ratio the students to the two groups extracted from the lists of students provided by the universities based on a table of random numbers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundamental of Care Framework implementation (Experimental): Educational interventions related to introduction of FoC framework and taking charge of patients and their fundamental needs will be realized during theoretical, simulation and internship learning.
  Interventions: Other: Theoretical and classroom learning interventions; Other: Simulation interventions; Other: Internship interventions
- No Fundamental of Care Framework implementation (No Intervention): the participants of no intervention group will receive the standard training as scheduled on the curriculum

INTERVENTIONS:
Other: Theoretical and classroom learning interventions — aim of intervention: introduce students to the conceptual framework of fundamental of care, focus on three dimensions necessary for the delivery of high-quality fundamental care (the nurse-patient relationship; addressing different fundamental needs; and a context that supports these goals)
  components and activities:
  * educational interventions to understand how the communication and the relationship of trust between nurse and patient are the prerequisites for high quality nursing care;
  * drawing attention to five essential relational elements for establishing the nurse-patient relationship (Trust; Focus; Anticipate; Know; Evaluate)
  mode of delivery:
  * classroom lessons on philosophies and theories on communication and trust
  * small-group learning on realistic cases focused on fundamental needs to develop reflexivity, analytical skills, investigation
  duration of the intervention: 12 hours of theoretical and classroom learning
  Arms: Fundamental of Care Framework implementation
Other: Simulation interventions — aim of intervention:
  To develop active listening and use of non-verbal and verbal communication skills to establish a therapeutic relationship based on compassion, trust and respect; to apply the FoC conceptual framework, reflexivity and analytical skills to meet patient fundamental needs.
  Students will express these goals during simulation activities with behaviours outlined by the FoC framework.
  components and activities: - Implementation of communication simulation activities to develop interaction skills with patients; Implementation of simulation activities to apply the FoC conceptual framework and reflection to meet patient fundamental needs in realistic scenarios.
  mode of delivery:
  - simulation activities on communication and trust Use ad hoc validated scenarios to apply the FoC conceptual framework to develop reflection and meet patient fundamental needs.
  duration of the intervention: 25 hours
  Arms: Fundamental of Care Framework implementation
Other: Internship interventions — Aim of intervention: to apply active listening and non-verbal communication skills; to use the FoC conceptual framework, reflexivity, and analytical skills to meet patient fundamental needs.
  Students will express these goals during simulation activities with behaviours outlined by the FoC framework.
  components and activities:
  - to establish effective and trusting communication with patients to demonstrate compassion and respect and to enable patients to remain calm, involved and dignified; to apply the FoC conceptual framework to meet patient fundamental needs.
  mode of delivery:
  * attendance of clinical internship
  * analysis and reflections guided by the clinical preceptor on real cases using elements of FoC conceptual framework.
  duration of the intervention: 150 hours of internship.
  Arms: Fundamental of Care Framework implementation

SUMMARY:
Research has shown a gap in what is important to patients and what is important to nurses when providing care. When the patient's fundamental needs are not recognized, such as hygiene, nutrition, mobilization, communication, he feels humiliated, ignored. The study aims to improve patient outcomes by educational interventions to integrate the Fundamental of Care (FoC) framework into nursing education.

A multi-centre randomized controlled trial will be conducted to evaluate the effectiveness of integrating the FoC framework into nursing education. Outcomes perceived by patients and their families relate to meeting the fundamental care needs.

DETAILED DESCRIPTION:
Background and Significance: Since 2010, to fill the gap in what is essential when providing care in a complex and challenging environment, both for patients and nurses, a line of research has developed to study the fundamental of nursing care. The "Fundamentals of Care (FoC) Frameworks" defines FoC as fundamental activities for the patient, through which the patient feels at the centre of care and feels attention and respect around him. The framework outlines three dimensions necessary for delivering high-quality fundamental care: the nurse-patient relationship; addressing different fundamental needs; and a context that supports these goals. A positive and trusting nurse-patient relationship is the basis for delivering fundamental care and forms the core of the framework.

FOCs are often implicit or invisible in nursing education, taught as an introductory part in the first year of the course and rarely addressed in subsequent years. The study aims to improve patient outcomes by educational interventions to integrate the FUNDAMENTAL OF CARE FRAMEWORK into nursing education.

Objectives: The substantive objectives of the study are: 1) To describe how nurses, internship preceptors, students and patients and their families perceive fundamental care; 2) Assessing learning process in developing FOC skills of nursing students; 3) Assessing nursing students perception of the learning environment and the supervision related to learning of FOC skills during the clinical internship; 4) Assessing the perceived outcomes of patients and their families related to meet the fundamental care needs.

Design: multi-centre randomized controlled trial

Sample: Students of nursing degree enrolled in the first year of the course, internship preceptors nurses who work in the internship departments of students enrolled in the first year of nursing degree, and patients over the age of 18, cognitively intact, assisted in the internship departments, who have the following three needs: (1) nutrition; (2) elimination; (3) personal hygiene will be included.

Measures: All outcomes will be measured with established criteria and with instruments used in previous studies or developed by the investigators and found validated and reliable.

Analysis: In addition to descriptive statistics, statistical tests to analyze differences in the scores between groups will be used to address the objectives.

ELIGIBILITY:
Inclusion Criteria:

* All students of nursing degree enrolled in the first year of the course who will choose to participate in the study
* All internship preceptors nurses who work in the internship departments of students enrolled in the first year of nursing degree will choose to participate in the study.
* All patients over the age of 18 assisted in the internship departments who choose to participate in the study who have the following three needs: (1) nutrition; (2) elimination; (3) personal hygiene.

Exclusion Criteria:

* Patients who are unable to answer the questionnaire independently, with altered mental status, with hospitalization of fewer than 24 hours

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
technical and relational FOC based performance of students after simulation. | At the end of simulation learning. (approximately 7 months after the beginning of the study)
  Technical and relational performance acquired on fundamental of care will be assessed by Objective Clinical Structured Examination (OSCE). Scenarios built ad hoc for applying the FoC conceptual framework will be used as an evaluation test. Checklists will be used for the assessment of technical skills and observation grids to assess communication skills.
  The student communication performance will be evaluated using a validated assessment grid (Guilbert, 1990), which consist of four variables (i.e., terminology, listening, attention, and clarity), broken down into five levels of expected, observable communicative behaviours. Values between -2 and +2 will be used to evaluate every variable.
  Checklists consist of a list of tasks. Each task will be evaluated with a score of 0 if not performed or performed incorrectly, with a score of 1 if performed correctly. The passing score is 80% of the tasks performed correctly.
technical and relational FOC based performance of students after internship. | At the end of internship learning. (approximately 10 months after the beginning of the study)
  Technical and relational performance acquired on fundamental of care will be assessed by Objective Clinical Structured Examination (OSCE). Scenarios built ad hoc for applying the FoC conceptual framework will be used as an evaluation test. Checklists will be used for the assessment of technical skills and observation grids to assess communication skills.
  The student communication performance will be evaluated using a validated assessment grid (Guilbert, 1990), which consist of four variables (i.e., terminology, listening, attention, and clarity), broken down into five levels of expected, observable communicative behaviours. Values between -2 and +2 will be used to evaluate every variable.
  Checklists consist of a list of tasks. Each task will be evaluated with a score of 0 if not performed or performed incorrectly, with a score of 1 if performed correctly. The passing score is 80% of the tasks performed correctly.

SECONDARY OUTCOMES:
Change of perception of fundamental of care by nurses, internship preceptors and students | perception of FoCs data will be collected at 3 time points: "baseline, before FoC framework training of trainers"; immediately after FoC framework training of trainers, immediately after the end of students' internship.
  All nurses working in the internship departments will be asked to answer the questionnaire that investigates how nurses perceive fundamental care concerning the importance, the frequency of implementation and the degree of responsibility perceived.
  The nursing perception questionnaire on fundamental nursing care consists of 4 sections (evaluation for every 13 fundamental needs in terms of importance recognized by organization and nurses, frequency of implementation, degree of responsibility perceived, need to have advanced competencies). The tool uses a five-point Likert scale and yes/no answers.
Change of perception of nursing students about how nursing student learn the fundamentals of care | Immediately after the end of students' theoretical, simulation and internship learning (complete FoC learning path). Approximately 10 months after the beginning of the study
  Skills acquired on fundamental of care will be assessed and how the learning process helps develop them by 'Fundamentals of Care' Learning Questionnaire - Basic Care Revised
  The questionnaire consists of 46 questions and uses a 4-point Likert scale to express the degree of agreement concerning learning fundamental of care and how it was learned (lesson or internship)
perception of nursing students on the learning environment and supervision of FOC learning during the clinical internship | Immediately after the end of students' internship (approximately 10 months after the beginning of the study)
  The Clinical Learning Environment, Supervision and Nurse Teacher Scale (CLES+T) scale consists of 34 statements divided into five sub-dimensions: "Pedagogical atmosphere on the ward" (nine items), "Leadership style of the ward manager" (four items), "Premises of nursing on the ward" (four items), "Supervisory relationship" (eight items) and "Role of the nurse teacher (NT)" (nine items). The CLES + T items are responded to on a 5-point Likert-type scale with higher values indicating more significant agreement with the statement.
perception of patients concerning to identification of fundamental needs and the responses received to these needs | During the students internship, at the end of hospitalization, immediately before discharge from the hospital (approximately 10 months after the beginning of the study)
  Patients will be asked to complete a questionnaire to evaluate:
  * the perception of fundamental needs present during the hospitalization;
  * identification of fundamental needs, indicated as being present by the patients, by the students during their internship;
  * effectiveness of interventions implemented by the clinical-care team to respond of fundamental needs indicated by patients The patient FoC outcomes questionnaire consists of 12 questions divided into five sub-dimensions: "Communication and education", "relationship", "Nutrition and hydration" , "Elimination" and "Personal hygiene and clothing" . The patient FoC outcomes items are responded to on a 4-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Bagnasco, Prof, Principal Investigator — Department of Health Sciences, University of Genoa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitson A, Conroy T, Wengstrom Y, Profetto-McGrath J, Robertson-Malt S. Defining the fundamentals of care. Int J Nurs Pract. 2010 Aug;16(4):423-34. doi: 10.1111/j.1440-172X.2010.01861.x. PMID 20649678
- [Background] Feo R, Kitson A. Promoting patient-centred fundamental care in acute healthcare systems. Int J Nurs Stud. 2016 May;57:1-11. doi: 10.1016/j.ijnurstu.2016.01.006. Epub 2016 Feb 1. PMID 27045560
- [Background] Bagnasco A, Timmins F, de Vries JMA, Aleo G, Zanini M, Catania G, Sasso L. Understanding and addressing missed care in clinical placements - Implications for nursing students and nurse educators. Nurse Educ Today. 2017 Sep;56:1-5. doi: 10.1016/j.nedt.2017.05.015. Epub 2017 May 23. PMID 28599196
- [Background] Feo R, Rasmussen P, Wiechula R, Conroy T, Kitson A. Developing effective and caring nurse-patient relationships. Nurs Stand. 2017 Mar 8;31(28):54-63. doi: 10.7748/ns.2017.e10735. PMID 28271761
- [Background] Feo R, Conroy T, Alderman J, Kitson A. Implementing fundamental care in clinical practice. Nurs Stand. 2017 Apr 5;31(32):52-62. doi: 10.7748/ns.2017.e10765. PMID 28378679
- [Background] Huisman-de Waal G, Feo R, Vermeulen H, Heinen M. Students' perspectives on basic nursing care education. J Clin Nurs. 2018 Jun;27(11-12):2450-2459. doi: 10.1111/jocn.14278. PMID 29399907
- [Background] Voldbjerg SL, Laugesen B, Bahnsen IB, Jorgensen L, Sorensen IM, Gronkjaer M, Sorensen EE. Integrating the fundamentals of care framework in baccalaureate nursing education: An example from a nursing school in Denmark. J Clin Nurs. 2018 Jun;27(11-12):2506-2515. doi: 10.1111/jocn.14354. PMID 29575165
- [Background] Saarikoski M, Warne T, Kaila P, Leino-Kilpi H. The role of the nurse teacher in clinical practice: an empirical study of Finnish student nurse experiences. Nurse Educ Today. 2009 Aug;29(6):595-600. doi: 10.1016/j.nedt.2009.01.005. Epub 2009 Feb 18. PMID 19232789
- [Derived] Bagnasco A, Lusignani M, Pagnucci N, Sallai T, Catania G, Napolitano F, Dal Molin A, Mazzoleni B, Cosmai S, Cattani D, Mansi L, Montani D, Zavaglio A, Sanvito P, Cartabia C, Consolo L, Giuseppe L, Zanini M, Sasso L. Italian Version of the Fundamentals of Care Framework and the Fundamentals of Care Practice Process: A Comprehensive Validation Study. J Adv Nurs. 2025 Jul 28. doi: 10.1111/jan.70099. Online ahead of print. PMID 40726058